CLINICAL TRIAL: NCT03482349
Title: A Prospective Randomized Clinical Trial (RCT) Comparing Functional and Radiographic Outcomes of Robotically-Assisted vs. Manually-Executed Total Knee Arthroplasties
Brief Title: RCT Comparing Robotically-Assisted vs. Manually-Executed Total Knee Arthroplasties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew P. Abdel, M.D., Associat Professor of Orthopedics, College of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-002188
Record Dates: First submitted 2018-02-15; First posted 2018-03-29 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total Knee Robotically-Assisted (Experimental): The intervention is then performed with a new device and surgical procedure. At first the femur and the tibia are fixed to the operating table with a special clamp and the knee bones are exposed with the standard technique; then the surgeon digitizes the shape of the joint and the computer transfers the planned surgical strategy to a dedicated surgical robot. Resections are performed by the surgeon on a constrained guide held by the robot.
  Interventions: Procedure: Total Knee Robotically-Assisted
- Total Knee Manual-Executed by Surgeon (No Intervention): Your orthopaedic surgeon will remove the damaged cartilage and bone, and then position the new metal and plastic implants to restore the alignment and function of your knee.

INTERVENTIONS:
Procedure: Total Knee Robotically-Assisted — The surgeon digitizes the shape of the joint and the computer transfers the planned surgical strategy to a dedicated surgical robot. Resections are performed by the surgeon on a constrained guide held by the robot.
  Arms: Total Knee Robotically-Assisted

SUMMARY:
This study will explore if there are any difference in functional outcomes between two different surgical procedures for total knee replacement: robot-assisted versus manually-executed total knee arthroplasty.

DETAILED DESCRIPTION:
Although total knee arthroplasty (TKA) is an effective treatment for end-stage knee arthritis, improvements in surgical technique remain a necessity. Contemporary designs have bolstered durability, but longer life expectancies have placed an even greater emphasis on survivorship. Additionally, patient satisfaction remains an issue.

A prospective randomized clinical trial (RCT) is proposed to compare robotically-assisted versus manually executed primary (TKAs). This study is designed to address the major short-term clinically important issues between the two types of procedures with special emphasis on functional outcome. Patients will be randomized to receive either a robotically-assisted or a manually-executed primary TKA.

ELIGIBILITY:
Inclusion Criteria:

* Include all patients who are surgical candidates for primary TKA with unilateral osteoarthritis
* All eligible male or female patients between the ages of 20 years to 100 years old
* All included study participants must be able to give an informed consent.

Exclusion Criteria:

* Significant femoral or tibial deformity due to congenital or traumatic etiologies, inflammatory arthritis, post-septic arthritis, osteomyelitis, prior infection of knee joint, osteoporosis, dislocated or fragmented patella
* The presence of infections, highly communicable diseases (e.g. AIDS), active tuberculosis, venereal disease, hepatitis.
* Significant neurological or musculoskeletal disorders or disease that may adversely affect normal gait or weight bearing.
* Presence of previous prosthetic knee replacement devices (of any type)
* Metastatic disease
* Psychiatric illness
* Drug or alcohol abuse
* Body mass index (BMI) > 40 kg/m2

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
Radiographic Parameters | 1 year
  Knee radiographs including an anteroposterior (AP) view and true lateral view, plus a patellar view

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P Abdel, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials